CLINICAL TRIAL: NCT06828393
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Single and Multiple Ascending Dose Trial of S-1117 in Healthy Volunteers
Brief Title: A Phase 1 Study of S-1117
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seismic Therapeutic AU Pty Ltd (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-1117-101
Record Dates: First submitted 2025-01-20; First posted 2025-02-14 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-1117 Part 1: Single ascending dose (SAD) cohorts (Experimental)
  Interventions: Drug: S-1117; Other: Placebo
- S-1117 Part 2: Multiple ascending dose (MAD) cohorts (Experimental)
  Interventions: Drug: S-1117; Other: Placebo

INTERVENTIONS:
Drug: S-1117 — S-1117 via subcutaneous or intravenous administration.
Other: Placebo — Placebo via subcutaneous or intravenous administration.

SUMMARY:
This is the first-in-human study of S-1117 designed to provide safety, tolerability, pharmacokinetic, and pharmacodynamic data in healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of S-1117 administered to healthy adult participants. This study will be conducted in two parts, Part 1 (single ascending dose, SAD) and Part 2 (multiple ascending doses, MAD).

ELIGIBILITY:
Major Inclusion Criteria:

1. Is available for the entire duration of the study and follow up.
2. Is willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.
3. Voluntarily consents to participation in the trial as documented by signing the study informed consent form (ICF).
4. Has a body mass index (BMI) within 18 to 32 kg/m2, inclusive, and weighs ≥45 kg.
5. Is in good physical and mental health in the opinion of the Investigator or delegate.

Major Exclusion Criteria:

1. Has a history of severe allergic or anaphylactic reaction as determined by the Investigator or delegate.
2. Is pregnant, nursing, or is planning to become pregnant or breastfeed during the trial.
3. Has a known immunodeficiency disorder.
4. Has a history of malignancy other than non-melanoma skin cancer.
5. Has a history of human immunodeficiency virus (HIV) or positive serology for HIV at Screening.
6. Has positive laboratory evidence for active hepatitis at screening.
7. Has received a live vaccine within 2 months of Screening.
8. Has any other condition or prior therapy that, in the opinion of the Investigator or delegate, may potentially compromise the safety or compliance of the participant, or may preclude the participant from successfully completing the study.

Other inclusion/exclusion eligibility criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse and serious adverse events as assessed by CTCAE v5.0 | 2 months

SECONDARY OUTCOMES:
To assess the maximum serum concentration (CMAX) | 2 months
To assess time to reach maximum serum concentration (tMAX) | 2 months
To assess elimination half-life (t1/2) | 2 months
To assess area under the serum concentration-time curve from time 0 to t hours (AUC0-t) and to infinity (AUC0-inf) | 2 months
To assess clearance (CL) | 2 months
To assess volume of distribution (Vz) and steady-state volume of distribution (Vss) | 2 months
To assess bioavailability after SC administration (F%) | 2 months
To characterize absolute and proportional change from baseline of immunoglobulin G (IgG) at multiple timepoints | 2 months
Incidence and characterization of antidrug antibody (ADA) | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Our IPD sharing plan is not yet developed. We will consider data sharing at a later date.